CLINICAL TRIAL: NCT04287855
Title: Multicenter Open Label Phase 2 Study of Isatuximab Plus Pomalidomide and Dexamethasone With Carfilzomib in Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Sanofi (Industry); Celgene (Industry); Amgen (Industry); Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IsKPd - IFM2018-03
Record Dates: First submitted 2020-01-31; First posted 2020-02-27 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; carfilzomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Isatuximab, Carfilzomib, Pomalidomide and Dexamethasone
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Isatuximab by IV route - Cycle 1 : 10mg/kg on days 1, 8, 15 and 22 per 28 days cycle. After cycle 1 : 10mg/kg on days 1 and 15 per 28 days cycle
Drug: Carfilzomib — Carfilzomib by IV route - Cycle 1 : 20/27 mg/m² on days 1-2, 8-9, 15-16 per 28 days cycle. Cycle 2-13 : 56mg/m² on days 1, 8, 15 per 28 days cycle. After cycle 13 : 56mg/m² on days 1 and 15 per 28 days cycle.
Drug: Pomalidomide — Pomalidomide by oral route - Cycle 1-2 : 3mg on days 1 to 21 per 28 days cycle. After cycle 2 : 4mg on days 1 to 21 per 28 days cycle.
Drug: Dexamethasone — Dexamethasone by oral route - Cycle 1-13 : 40/20 mg on days 1, 8, 15 and 22. Cycle 2-13 : 56mg/m² on days 1, 8, 15 per 28 days cycle. After cycle 13 : 56mg/m² on days 1 and 15 per 28 days cycle.

SUMMARY:
Study a quadruplet-based regimen with Minimal Residual Disease (MRD) 10-5 negative rate as primary end point in patients with early Relapsed or Refractory Multiple Myeloma.

Therapeutic study, phase II, prospective, multicenter, open-label. The patients will be treated until progression. Each cycle of treatment lasts 28 days. Cycle 1 to 13 : treatment phase After cycle 13 : maintenance phase

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and voluntarily sign an informed consent form
2. Must be able to adhere to the study visit schedule and other protocol requirements
3. Male or female, age 18 years or older
4. Life expectancy of > 6 months.
5. Must have a in R1 and R2 relapse Multiple Myeloma with a measurable disease :

   * 1 to maximum 2 lines of therapy prior to study entry
   * Relapse Refractory or primary refractory or relapse
   * Must have received prior treatment with a Lenalidomide-containing regimen for at least 2 consecutive cycles
6. Must have measurable disease as defined by the following: must have a clearly detectable and quantifiable monoclonal M-component value in the serum and/or urine :

   * IgG/IgA (serum M-component > 5g/l),
   * Light chain (serum M-component >1g/l or Bence Jones > 200mg/24H),
   * Serum FLC assay (including for IgD isotypes): involved FLC level > 10 mg/dl provided serum.

   FLC ratio is abnormal for patients not measurable on any of the 3 above criteria.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
8. Wash out period without MM treatment must be of 28 days minimum before C1D1, except for anti CD-38 (See exclusion criteria#10).
9. Adequate bone marrow function, documented within 72 hours and without transfusion 72 hours prior to the first intake of investigational product (C1J1) with no growth factor support (one week), defined as :

   * Absolute neutrophils ≥ 1 x109/L,
   * Untransfused Platelet count ≥ 75 x109/L,
   * Hemoglobin ≥ 8.5 g/dL.
10. Adequate organ function defined as :

    * Serum total bilirubin < 2x upper limit of normal (ULN),
    * Clearance creatinine ≥ 30ml/min,
    * Serum SGOT/AST or SGPT/ALT < 3x upper limit of normal (ULN).
11. Patients affiliated to an appropriate social security system.
12. A man who is sexually active with a pregnant female or a FCBP* must agree to use a barrier method of birth control eg, condom with spermicidal foam/gel/film/cream/suppository, even if he has had a vasectomy. All men must also not donate sperm, spermatozoa during the study, for 5 months following treatment discontinuation.
13. A woman FCBP* must understand and agree to use 2 reliable effective methods (a very effective method and an effective additional method) of contraception simultaneously without interruption :

    * For at least 28 days before starting experimental treatments,
    * Throughout the entire duration of experimental treatments,
    * During dose interruptions,
    * And for at least 5 months after the last dose of experimental treatments.
14. All patients must agree to not donate blood during the treatment period, interruptions of treatment and at least 5 months after the last dose of treatment.
15. All patients must understand and accept to comply with the conditions of the Pomalidomide pregnancy prevention plan (Appendix of the protocol).

Exclusion Criteria:

1. Any other uncontrolled medical condition or comorbidity that might interfere with patient's participation, including simultaneous participation to another interventional clinical study.
2. Known positive for HIV or active infectious hepatitis, type B or C.
3. Patients with non-secretory MM and non-measurable MM
4. Patient with terminal renal failure that require dialysis or clearance creatinine < 30 ml/min (calculated with MDRD formula)
5. Any uncontrolled or severe cardiovascular or pulmonary disease determined by the investigator including :

   * NYHA functional classification III or IV congestive heart failure
   * LVEF (Left Ventricular Ejection Fraction) < 40%
   * Uncontrolled angina, hypertension or arrhythmia
   * Myocardial infarction in the past 6 months
6. Prior history of malignancies, other than multiple myeloma, unless the patients has been free of the disease for ≥ 5 years. Exceptions include the following:

   * Basal or squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix or breast
   * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
7. Evidence of central nervous system (CNS) involvement
8. Ongoing active infection or other clinically significant uncontrolled cardiovascular events
9. Unable to comply with IMids regulation to thromboprophylaxis, or teratogenic recommandations.
10. Refractory to prior to anti CD38.Patients can be exposed to anti CD38 (any), BUT the wash out period for patient pre-treated with an anti CD38 antibody must be of 4,5 months minimum between last dose of previous anti-CD38 antibody and the first dose of isatuximab.
11. Refractory to prior carfilzomib
12. Known allergy to one of the study product (pomalidomide, isatuximab, carfilzomib) or dexamethasone
13. Patient with a history of severe allergic reactions to thalidomide or lenalidomide
14. Exposed to pomalidomide
15. Known intolerance to infused protein products, sucrose, histidine, and PS80
16. Contraindications to dexamethasone
17. Any ongoing non hematological adverse event or medical history grade> 2 severity
18. Pregnant or breast-feeding females
19. Refusal to participate in the study
20. Persons protected by a legal regime (guardianship, trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of trial treatment | Up to 5 years
  Fraction of patients who experience a Minimal Residual Disease (MRD) 10-5 per IMWG (International Myeloma Working Group) criteria

SECONDARY OUTCOMES:
Safety of trial treatment | Up to 5 years
  List of AE frequency (AE assessed by Common Terminology Criteria for Adverse Events (CTCAE) criteria, version 5.0)
Depth of response to the trial treatment | Up to 5 years
  Per International Myeloma Working Group (IMWG) criteria
Progression Free survival | Up to 5 years
  Time to relapse or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: LELEU Xavier, Prof., Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU Poitiers, Poitiers, France